CLINICAL TRIAL: NCT02930408
Title: Compare Train and 3D-4D Left Ventricular Systolic Function in Subjects Suffering From Dystrophy and Healthy Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: STEINECHO
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-08

CONDITIONS: Steinert's Disease
MeSH Terms: conditions — Myotonic Dystrophy

INTERVENTIONS:
Procedure: electrocardiogram
Procedure: Echocardiography

SUMMARY:
Steinert's disease is an orphan disease. The prognosis of patients with this disease is conditioned by cardiac involvement. Search an early stage alterations in contractile function in subjects suffering from dystrophy would detect patients at risk of sudden death. The first stage of work is to validate the tools to detect early stage of infringement systolic function in a population of patients with myotonic dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from muscular dystrophy type 1 followed CHU Poitiers.
* age ≥ 18 years

Exclusion Criteria:

* duration QRS> 120 ms ECG permanent ventricular stimulation
* trouble segmental kinetic obvious to echocardiography in visual analysis

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Ventricular Ejection Fraction Left 3D | Immediately
Global longitudinal systolic Strain | Immediately
Strain of the dispersion index | Immediately